CLINICAL TRIAL: NCT02882893
Title: Efficacy and Safety of DWP450 for the Treatment of Crows Feet Lines: Active Controlled, Double-blind, Randomized, Multi-center, Phase II/III Clinical Trial
Brief Title: Efficacy and Safety of DWP450 for the Treatment of Crows Feet Lines
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP450005
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Crows Feet Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DWP450 (Experimental): Single-dose
  Interventions: Drug: Clostridium Botulinum A Toxin
- Botox (Active Comparator): Single-dose
  Interventions: Drug: Clostridium Botulinum A Toxin

INTERVENTIONS:
Drug: Clostridium Botulinum A Toxin
  Other Names: BOTOX
  Arms: Botox
Drug: Clostridium Botulinum A Toxin
  Other Names: NABOTA
  Arms: DWP450

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of DWP450 treatment of Crows Feet Lines(CFL).

ELIGIBILITY:
Inclusion Criteria:

* Male or female of at least 18 to 75 years old
* Bilaterally symmetrical moderate-to-severe CFL at maximum smile on the FWS as rated by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Facial Wrinkle Scale(FWS) severity of Crow's feet lines(CFL) at maximum smile as assessed by investigators | At 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No